CLINICAL TRIAL: NCT03917641
Title: Effectiveness of Khat on Eyelid Wound Healing After Oculoplastic Surgery - a Prospective Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-17-4804-GBS-CTIL
Record Dates: First submitted 2019-04-01; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hematoma; Surgical Wound; Surgery; Eye Bruise; Edema
Keywords: Oculoplastic Surgery; Khat leaves; Post operative care; Edema; Hematoma
MeSH Terms: conditions — Hematoma; Surgical Wound; Edema

STUDY DESIGN:
Intervention Model Description: Each participant is his own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients after Oculoplastic surgery (Experimental): Each participant will use one compression with Khat leaves and another standard compression and will decide on which eye to use which compression.
  The compressions will be used for 10 minutes per every waking hour in the first 2 days post-op.
  The patient will take pictures of both his eyes in days 1,3 and 7 post operative days.
  Interventions: Biological: Khat leaves

INTERVENTIONS:
Biological: Khat leaves — One of the two compressions (one per each eye) the patient will use will contain the Khat leaves.

SUMMARY:
The post operative routine after Oculoplastic Surgery includes usage of cold compressions for symptomatic relief and decreasing of the edema and local hematomas in the first few days after the surgery. Khat (Catha edulis) is a plant that is used mainly for chewing and has a known stimulating effect, some patients report major improvement after including these leaves in the compressions they use after surgery. Khat contains the chemical ingredients Cathine and Cathinone, which are amphetamine-like alkaloids and probably the main contributors for its active effects. Our main goal is to use compressions that include the Khat leaves and check their effect on reducing the edema and hematomas after oculoplastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent blepharoplasty and/or ptosis repair

Exclusion Criteria:

* Patients who were operated on one eye only
* Patients who underwent a different surgery in each eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Edema | 7 days post op
  Improvement in edema in the Khat compression in comparison to standard compression by clinical evaluation.
Hematoma | 7 days post op
  Improvement in hematomas in the Khat compression in comparison to standard by compression by clinical evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malhotra R, Ziahosseini K, Poitelea C, Litwin A, Sagili S. Effect of Manuka Honey on Eyelid Wound Healing: A Randomized Controlled Trial. Ophthalmic Plast Reconstr Surg. 2017 Jul/Aug;33(4):268-272. doi: 10.1097/IOP.0000000000000743. PMID 27429228